CLINICAL TRIAL: NCT07238894
Title: Peking University People's Hospital Breast Surgery Department
Brief Title: A Cohort Study of Combined Cryoablation and Thermal Ablation for Non-surgical Treatment of Breast Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Shu Wang, director of breast center, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUPHBC202509
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Ablation; Breast Cancer
Keywords: Combined Cryoablation and Thermal Ablation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined Cryoablation and Thermal Ablation for Non-surgical Treatment of Breast Cancer Patients (Experimental)
  Interventions: Device: Combined Cryoablation and Thermal Ablation system

INTERVENTIONS:
Device: Combined Cryoablation and Thermal Ablation system — The combined cold and heat ablation system, as an advanced minimally invasive medical device for tumors independently developed in China, adopts a combined mode of deep low-temperature cryotherapy and high-intensity heating to treat tumors. This system uses liquid nitrogen as the refrigerant, which is easy to obtain. The minimum freezing temperature can reach -196℃, and the single-needle ablation range is larger. Using anhydrous ethanol as the heat medium, the ablation needle can be heated to 80℃ after freezing, which can dissolve ice balls more quickly. At the same time, it can ablate the puncture needle tract, reduce bleeding, prevent tumor needle tract implantation and metastasis, and has higher safety.

SUMMARY:
Although surgical resection is the gold standard for early breast cancer treatment, some patients cannot tolerate surgery due to medical conditions or refuse surgical treatment for cosmetic reasons. In recent years, the rapid development of ablation technology has provided new directions for breast cancer patients who are not suitable for surgical treatment. Ablation uses high or low temperatures to deactivate lesions or tissues, which are gradually absorbed by the body, achieving local treatment purposes. Its safety and efficacy have been preliminarily confirmed. As an advanced minimally invasive medical device independently developed in China, the combined cryo-thermal ablation system treats tumors using a combined mode of deep cryogenic freezing and high-intensity heating. It has been approved for ablation treatment of various solid tumors including lung cancer, pancreatic cancer, kidney cancer, prostate cancer, breast cancer, bone and soft tissue sarcomas.

This project proposes a prospective cohort design, based on the breast disease cohort database of Peking University People's Hospital Breast Center. It will enroll patients pathologically diagnosed with breast cancer, determined unsuitable for surgical treatment, and have received combined cryo-thermal ablation. The registered data will be used to evaluate the effectiveness and safety of percutaneous ultrasound-guided cryo-thermal composite ablation in this population.

DETAILED DESCRIPTION:
1. Study Design

1. Prospective Cohort Study Study Subjects and Selection Criteria
2. This study is based on the breast disease cohort database of Peking University People's Hospital Breast Center. Patients with pathologically confirmed breast cancer who refused, were intolerant of, or unsuitable for surgical treatment and received combined cryoablation and thermal ablation were prospectively enrolled.

The specific inclusion and exclusion criteria are as follows:

1. Inclusion Criteria (all conditions must be met):

   ≥18 years old; Breast cancer confirmed by core needle biopsy; Tumor lesions clearly visible on ultrasound; No contraindications for cryoablation such as coagulation disorders;

   Presence of reasons unsuitable for conventional surgical resection:

   Patients intolerant to general anesthesia or surgical treatment due to medical conditions; Due to unresectable and/or metastatic disease; Patient refusal of surgery, etc.; Agree to undergo ablation surgery and sign the informed consent form.
2. Exclusion Criteria (Participants will be excluded if any of the following apply):

Missing clinical and pathological data (such as imaging or pathological materials); Pregnant or lactating women; Known allergies, intolerance, or contraindications to cryotherapy (such as cryoglobulinemia, presence of implanted electronic devices); Vulnerable populations, including those with neurological disorders, cognitive impairments, critically ill patients, etc.

3)Grouping of Study Subjects This study is a prospective cohort study. The decision to undergo combined cold and heat ablation therapy was made through mutual consultation between patients and attending physicians, while the remaining systemic treatments were not affected by the study.Cohort 1: Ablation therapy for patients who cannot tolerate standard surgery due to advanced age or comorbidities;Cohort 2: Ablation therapy for patients with unresectable/metastatic diseases who are not suitable for surgical resection;Cohort 3: Ablation therapy chosen by patients who refuse surgical treatment for personal reasons.

4)Research Steps Screen patients who meet the inclusion criteria and exclude those who meet the exclusion criteria.

Collect patients' clinicopathological data: age, menstrual status, accompanying diseases; tumor imaging information, including ultrasound, mammography, MRI reports, tumor size, and axillary lymph node status; pathological information, including pathological type, histological grade, hormone receptor status, and postoperative adjuvant treatment plans.

Breast primary tumors receive standard combined cryoablation and thermal ablation treatment, and collect imaging and histological laboratory data during and after treatment.

Retrieve patients' prognosis information from the follow-up database, including recurrence, metastasis, second primary tumor, and mortality events.

5)Follow-up Plan and Contents:

Postoperative Complications (within 3 months):

Skin damage Poor incision healing Infection Seroma formation Nipple or flap ischemia/necrosis

Survival-related Follow-up:

Recurrence Metastasis Second primary tumor Mortality events

Follow-up Methods:

Telephone WeChat client of Peking University People's Hospital Follow-up System Follow-up Interval: 6 months Follow-up Duration: More than 5 years 6)Selection and Confirmation of Primary Measurement Indicators or Outcome Measures

Primary Study Endpoint - Safety:

Intraoperative complications (e.g., bleeding, vascular/nerve injury) Postoperative complications (infection, hematoma, frostbite, breast deformity, paresthesia, etc.), recorded according to CTCAE v5.0 classification Local tumor recurrence rate (Ipsilateral Breast Cancer Recurrence, IBTR): defined as the time from surgery to ipsilateral breast tumor recurrence, with the occurrence of ipsilateral breast tumor recurrence as the event

Secondary Study Endpoints:

Disease-free survival (DFS): time from study enrollment to the first occurrence of failure events, including ipsilateral local-regional recurrence, contralateral breast cancer, distant recurrence, or death from any cause Overall survival (OS): time from study enrollment to death from any cause Exploratory analysis: using specimen bank preserved samples and imaging data to analyze post-ablation tumor tissue pathological response, blood immune function assessment, and the correlation between postoperative imaging (MRI/ultrasound) characteristics and recurrence risk All data collection is sourced from the established Peking University People's Hospital Breast Disease Cohort Database (PKUPH Breast Disease Cohort).

7)The primary study outcome was a local IBTR at 5 years through the width of the 95% conﬁdence interval (CI). A sample size was calculated for this outcome. For a two-sided 95% exact Clopper Pearson conﬁdence interval of the IBTR rate whose true value was 5%, a sample size of 200 patients was required to yield a half-width of 5% at most with more than 99% power. In this context, power is the probability (conditional method) of obtaining a conﬁdence interval a half-width less than or equal to the hypothesized value.

ELIGIBILITY:
Inclusion Criteria:

* 1) Aged 18 or above; 2) Breast cancer confirmed by core needle biopsy; 3) Tumor lesions clearly visible on ultrasound; 4) No contraindications for cryoablation such as coagulation disorders; 5) Presence of reasons unsuitable for conventional surgical resection: patient's condition cannot tolerate general anesthesia or surgical treatment; due to unresectable and/or metastatic disease; patient refuses surgery, etc.; 6) Agree to undergo ablation surgery and sign the consent form.

Exclusion Criteria:

* 1) Missing clinical and pathological data (such as imaging and pathological materials); 2) Pregnant or lactating women; 3) Known allergies, intolerances, or contraindications to cryotherapy (such as cryoglobulinemia, presence of implanted electronic devices); 4) Vulnerable populations, including those with neurological disorders, cognitive impairments, critically ill patients, etc.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer patient
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Ipsilateral breast cancer recurrence | 3 years
  From the surgery date to the ipsilateral breast tumor recurrence date
the rate of comlications | 3 months
  The proportion of complications occurring during surgery and within 3 months after surgery

SECONDARY OUTCOMES:
disease free survival | 3 years
  The time from enrollment to the first occurrence of the following events defined as failure, including ipsilateral local recurrence, contralateral breast cancer, distant recurrence or death from any cause.
overall survival | 3 years
  The time from enrollment to death caused by any reason.

OTHER OUTCOMES:
exploratory research | 1 year
  Correlation analysis between pathological reactions of tumor tissue after ablation, evaluation of blood immune function, postoperative imaging (MRI/ultrasound) features and recurrence risk, etc

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Yang W, An Y, Li Q, Liu C, Zhu B, Huang Q, Zhao M, Yang F, Feng H, Hu K. Co-ablation versus cryoablation for the treatment of stage III-IV non-small cell lung cancer: A prospective, noninferiority, randomized, controlled trial (RCT). Thorac Cancer. 2021 Feb;12(4):475-483. doi: 10.1111/1759-7714.13779. Epub 2020 Dec 14. PMID 33319493
- [Result] Wang YF, Li XG. Co-ablation of lung malignancies with coexisting usual interstitial pneumonia: a retrospective analysis of safety and efficacy. Int J Hyperthermia. 2025 Dec;42(1):2468764. doi: 10.1080/02656736.2025.2468764. Epub 2025 Feb 23. PMID 39988332
- [Result] Fine RE, Gilmore RC, Tomkovich KR, Dietz JR, Berry MP, Hernandez LE, Columbus KS, Seedman SA, Fisher CS, Han LK, Manahan ER, Hicks RD, Vaidya RP, Curcio LD, Sevrukov AB, Kenler AS, Taback B, Chen M, Miller ME, Gold L, Anglin BV, Aoun HD, Simmons RM, Feldman SM, Boolbol SK. Cryoablation Without Excision for Early-Stage Breast Cancer: ICE3 Trial 5-Year Follow-Up on Ipsilateral Breast Tumor Recurrence. Ann Surg Oncol. 2024 Oct;31(11):7273-7283. doi: 10.1245/s10434-024-16181-0. Epub 2024 Sep 16. PMID 39283572
- [Result] Fine RE, Gilmore RC, Dietz JR, Boolbol SK, Berry MP, Han LK, Kenler AS, Sabel M, Tomkovich KR, VanderWalde NA, Chen M, Columbus KS, Curcio LD, Feldman SM, Gold L, Hernandez L, Manahan ER, Seedman SA, Vaidya RP, Sevrukov AB, Aoun HD, Hicks RD, Simmons RM. Cryoablation Without Excision for Low-Risk Early-Stage Breast Cancer: 3-Year Interim Analysis of Ipsilateral Breast Tumor Recurrence in the ICE3 Trial. Ann Surg Oncol. 2021 Oct;28(10):5525-5534. doi: 10.1245/s10434-021-10501-4. Epub 2021 Aug 15. PMID 34392462
- [Result] van de Voort EMF, Struik GM, Birnie E, Moelker A, Verhoef C, Klem TMAL. Thermal Ablation as an Alternative for Surgical Resection of Small (</= 2 cm) Breast Cancers: A Meta-Analysis. Clin Breast Cancer. 2021 Dec;21(6):e715-e730. doi: 10.1016/j.clbc.2021.03.004. Epub 2021 Mar 17. PMID 33840627
- [Result] Wang YQ, Tan ZK, Peng Z, Huang H. A systematic review and meta-analysis of the comparison of laparoscopic radiofrequency ablation to percutaneous radiofrequency ablation for hepatocellular carcinoma. Front Oncol. 2025 Mar 11;15:1559343. doi: 10.3389/fonc.2025.1559343. eCollection 2025. PMID 40134600
- [Result] Azizi M, Heshmatnia F, Milani H, Shahhosseini Z, Marvdashti LM, Moghadam ZB. The Effectiveness of Cognitive Behavioral Therapy on Depression and Anxiety Symptoms in Breast Cancer Patients and Survivors: A Systematic Review of Interventional Studies. Brain Behav. 2024 Oct;14(10):e70098. doi: 10.1002/brb3.70098. PMID 39467209
- [Result] Divani A, Heidari ME, Ghavampour N, Parouhan A, Ahmadi S, Narimani Charan O, Shahsavari H. Effect of cancer treatment on sleep quality in cancer patients: A systematic review and meta-analysis of Pittsburgh Sleep Quality Index. Support Care Cancer. 2022 Jun;30(6):4687-4697. doi: 10.1007/s00520-021-06767-9. Epub 2022 Jan 26. PMID 35079904
- [Result] Ziegler P, Hartkopf AD, Wallwiener M, Haberle L, Kolberg HC, Hadji P, Tesch H, Ettl J, Luftner D, Muller V, Michel LL, Belleville E, Wimberger P, Hielscher C, Huebner H, Uhrig S, Wurmthaler LA, Hack CC, Mundhenke C, Kurbacher C, Fasching PA, Wuerstlein R, Untch M, Janni W, Taran FA, Lux MP, Wallwiener D, Brucker SY, Fehm TN, Schneeweiss A, Goossens C. The impact of physical activity on progression-free and overall survival in metastatic breast cancer based on molecular subtype. BMC Cancer. 2024 Oct 16;24(1):1284. doi: 10.1186/s12885-024-13038-3. PMID 39415149
- [Result] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Kim J, Harper A, McCormack V, Sung H, Houssami N, Morgan E, Mutebi M, Garvey G, Soerjomataram I, Fidler-Benaoudia MM. Global patterns and trends in breast cancer incidence and mortality across 185 countries. Nat Med. 2025 Apr;31(4):1154-1162. doi: 10.1038/s41591-025-03502-3. Epub 2025 Feb 24. PMID 39994475